CLINICAL TRIAL: NCT01933269
Title: Initial Evaluation of Anti-1-amino-F-18 Flurocyclobutane-1carboxylic Acid (Anti-18F-FACBC) in the Assessment of Head and Neck Cancer: A Pilot Study.
Brief Title: FACBC for Head and Neck Cancers
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Change in Principal Investigator and protocol revisions delayed study start and ultimately the decision was made to cancel the study.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David M. Schuster, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00062214
Record Dates: First submitted 2013-08-16; First posted 2013-09-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cancers of the Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FACBC (Experimental)
  Interventions: Drug: FACBC

INTERVENTIONS:
Drug: FACBC

SUMMARY:
The purpose of this study is to assess a relatively new PET (Positron emission tomography) radiotracer called FACBC in the assessment of head and neck cancer. FDG (Flourine Deoxyglucose) is currently used for PET imaging, but has limitations in head and neck cancer. These limitations include problems with specificity, high background uptake from normal structures, difficulty delineating intracranial invasion, and the need to wait several weeks after chemotherapy and radiation before imaging. As an amino acid radiotracer, rather than a glucose radiotracer, FACBC overcomes some of these limitations. FACBC does not yet have FDA (Food and Drug Administration) approval, but does show promise in initial work in patients with prostate cancer and brain tumors. Dosimetry work on FACBC has been performed at Emory.

Our study is a pilot study looking at 10 patients with a new diagnosis of biopsy proven squamous cell carcinoma of the oral cavity who will be able to go on to definitive surgical resection (ie, surgery without preceding chemotherapy or radiation). Patients must have pre-surgical imaging, either with a contrast enhanced CT, FDG PET, or MRI. Patients who consent to participate will receive one FACBC PET/CT of the neck, which will require a low dose "transmission" CT of the neck, an intravenous injection of the radiotracer, and imaging of the neck that will last up to 1 hour. Patients will have to lie still during the imaging time. Total participation time including set up should be less than 90 minutes. Imaging results will be analyzed and compared with conventional imaging as well as the surgical pathology results

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Biopsy proven, untreated squamous cell carcinoma of the oral cavity.
3. Clinical, laboratory, or diagnostic imaging findings on CT, MRI, or 18F-FDG PET/CT.
4. Ability to lie still for PET scanning.
5. Able to provide written informed consent.

Exclusion Criteria:

1. Age less than 18 years.
2. Prior history of carcinoma.
3. Not a candidate for surgical resection based upon clinical condition or discovery of metastatic disease which would preclude surgical therapy.
4. Inability to lie still for PET scanning.
5. Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
The presence of FACBC radiotracer uptake in Head and neck tumors on PET scans | 1 day
  The results of the FACBC PET scan will be validated by direct comparison with the pathology findings obtained at surgery. .

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Karagulle Kendi, MD, Principal Investigator — Emory University; David Schuster, MD, Study Director — Emory University